CLINICAL TRIAL: NCT03495921
Title: A Multi-Center Phase III, Randomized, Open-Label Trial of Vigil (Bi-shRNAfurin and GMCSF Augmented Autologous Tumor Cell Immunotherapy) in Combination With Irinotecan and Temozolomide as a Second-Line Regimen for Ewing's Sarcoma
Brief Title: A Trial For Participants With Ewing's Sarcoma Treated With Vigil in Combination With Irinotecan and Temozolomide
Acronym: VITA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow accrual and as a result, a strategic business decision was made to terminate enrollment.
Sponsor: Gradalis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL-PTL-130
Expanded Access: NCT03842865 (Temporarily not available)
Record Dates: First submitted 2018-02-15; First posted 2018-04-12 (Actual); Results first posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Ewing Sarcoma; Ewing Family of Tumors; Ewing's Tumor Metastatic; Ewing's Sarcoma Metastatic; Ewing's Tumor Recurrent; Rare Diseases; Sarcoma; Neoplasms, Connective and Soft Tissue; Neoplasms by Histologic Type; Neoplasms, Bone Tissue; Neoplasms, Connective Tissue; Sarcoma, Ewing; Neoplasms
Keywords: ESFT; Immunotherapy; Phase 3; irinotecan; temozolomide; First Relapse; Second Line; Vigil; vaccine; orphan drug; soft bone; pediatric; FLI; EWS; Molecular Mechanisms of Pharmacological Action; Antineoplastic Agents
MeSH Terms: conditions — Sarcoma, Ewing; Neuroectodermal Tumors, Primitive, Peripheral; Rare Diseases; Sarcoma; Neoplasms, Connective and Soft Tissue; Neoplasms by Histologic Type; Neoplasms, Bone Tissue; Neoplasms, Connective Tissue; Neoplasms | interventions — FANG vaccine; Irinotecan; Temozolomide

STUDY DESIGN:
Intervention Model Description: Participants were randomized 1:1 to either Group A (Vigil + irinotecan and temozolomide) or Group B (irinotecan and temozolomide alone). Participants randomized to Group B were able to receive Vigil (Cross-Over) after confirmation of progression by central radiologist and sponsor approval.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group A: Vigil + Irinotecan and Temozolomide (Experimental): Participants randomized to Group A received oral temozolomide 100 mg/m2 daily (Days 1-5), total dose 500 mg/m2/cycle) and oral irinotecan 50 mg/m2 daily (Days 1-5, total dose 250 mg/m2/cycle). Vigil immunotherapy was administered at a concentration of 1 X 10e6 cells/dose given via intradermal injection on Day 15 of each cycle. 1 cycle = 21 days
  Participants continued treatment for a maximum of 12 cycles, or until disease progression, unacceptable toxicity, withdrawal of consent or other criterion is met for discontinuation from study.
  Interventions: Biological: Vigil; Drug: Irinotecan; Drug: Temozolomide
- Group B: Irinotecan and Temozolomide (Active Comparator): Participants randomized to Group B received oral temozolomide 100 mg/m2 daily (Days 1-5), total dose 500 mg/m2/cycle) and oral irinotecan 50 mg/m2 daily (Days 1-5, total dose 250 mg/m2/cycle).
  1 cycle = 21 days
  Participants continued treatment for a maximum of 12 cycles, or until disease progression, unacceptable toxicity, withdrawal of consent or other criterion is met for discontinuation from study.
  Interventions: Drug: Irinotecan; Drug: Temozolomide
- Cross-Over: Vigil monotherapy (Other): Participants randomized to Group B were able to receive Vigil immunotherapy at a concentration of 1 X 10e6 cells/dose given via intradermal injection on Day 15 of each cycle. Confirmation of progression by central radiologist and pre-approval from sponsor was required. 1 cycle = 21 days
  Interventions: Biological: Vigil

INTERVENTIONS:
Biological: Vigil — Vigil is composed of autologous tumor cells harvested from the patient at the time of initial de-bulking surgery which are then transfected extracorporeally, with a plasmid encoding for the gene for GM-CSF, an immune-stimulatory cytokine, and a bifunctional, short hairpin RNA which specifically knocks down the expression of furin, the critical convertase responsible for production of the two TGβ isoforms.
  Other Names: Bi-shRNAfurin and GMCSF Augmented Autologous Tumor Cell Immunotherapy; FANG vaccine
  Arms: Cross-Over: Vigil monotherapy; Group A: Vigil + Irinotecan and Temozolomide
Drug: Irinotecan — Injectable formulation of irinotecan was distributed from central supplier. 1 Cycle (5 doses of 50 mg/m2 per syringe) was drawn into provided oral syringes and dispenses to the subject with instructions to refrigerate until administration.
  Other Names: Camptosar; Camptothecin-11; CPT-11
  Arms: Group A: Vigil + Irinotecan and Temozolomide; Group B: Irinotecan and Temozolomide
Drug: Temozolomide — Dose: 100 mg/m2 daily, oral Schedule: Days 1-5, every 21 days Administered at least 1 hour before Irinotecan.
  Other Names: Temodar
  Arms: Group A: Vigil + Irinotecan and Temozolomide; Group B: Irinotecan and Temozolomide

SUMMARY:
The goal of this clinical trial was to compare participants with first relapse or refractory Ewing's sarcoma when treated with investigational product (Vigil) in addition to the standard treatment of irinotecan and temozolomide compared to the standard treatment of irinotecan and temozolomide alone. The main question it aimed to answer is "Will participants who receive Vigil in addition to irinotecan and temozolomide have a prolonged time to progression and improved quality of life compared to the participants who receive irinotecan and temozolomide alone?".

DETAILED DESCRIPTION:
This was a multicenter, Phase III study in participants with metastatic Ewing's sarcoma Family of Tumors (ESFT) refractory/intolerant or recurrent to 1 prior line of chemotherapy. Participants who agreed to participation had tumor tissue harvested from a scheduled standard surgical procedure (e.g., tumor biopsy or palliative resection). The tumor tissue removed was shipped to Gradalis, Inc. to attempt to manufacture the investigational product, Vigil.

Subjects who met eligibility criteria including manufacture of a minimum of 4 doses of Vigil were randomized 1:1 to either Group A (Vigil + Irinotecan + Temozolomide (Tem/Iri)) or Group B (Irinotecan + Temozolomide). Screening for the main portion of the study occurred as early as one week but no later than 8 weeks following tumor procurement.

Subjects received repeat cycles of treatment until disease progression, unacceptable toxicity, withdrawal of consent or other criterion was met for discontinuation from study. Subjects randomized to Group A (Vigil + Tem/Iri) received up to 12 doses depending upon the quantity of Vigil manufactured from the surgical specimen. 1 cycle = 21 days. If irinotecan + temozolomide was administered beyond 12 cycles, it was administered off study. Subjects randomized to Group B (Tem/Iri) may have crossed over to receive single agent Vigil every 21 days following End of Treatment assessment and documented disease progression confirmed by central radiology vendor, for up to 12 doses of Vigil depending upon the quantity of Vigil manufactured.

Participants were managed in an outpatient setting. Hematologic function, liver enzymes, renal function and electrolytes will be monitored. Blood for immune function analyses including IFNγ-ELISPOT analysis of cytotoxic T cell activation in response to autologous tumor antigens will be collected at tissue procurement, post-procurement screening and Day 1 (prior to chemotherapy administration) at Cycles 2, 4, and 6, end of treatment (EOT), 3 months after EOT, and every 6 months thereafter. Blood for ctDNA analysis was collected at tissue procurement, prior to chemotherapy administration at baseline and on Day 1 prior to chemotherapy administration at Cycles 2, 3, 4, and 6, and EOT. After progression, participants were contacted quarterly for documentation of post study therapies and survival status information.

ELIGIBILITY:
Tissue Procurement Inclusion Criteria:

1. Histologically confirmed Ewing's Sarcoma Family of Tumors (ESFT).
2. Age greater than or equal to 2 years.
3. Estimated survival greater than or equal to 6 months.
4. Evidence of EWS translocation by FISH or RT-PCR or Next Generation Sequencing (NGS). If available, NGS sequencing report should be submitted to Gradalis.
5. Recurrence or refractory to 1 line of systemic chemotherapy, including but not limited to doxorubicin, vincristine, and ifosfamide.
6. Planned standard of care surgical procedure (e.g., tumor biopsy or palliative resection or thoracentesis) and expected availability of a cumulative soft-tissue mass of ~10-30 grams tissue ("grape" to "golf-ball" size / approximately 2 cm total diameter on imaging) or pleural fluid estimated volume ≥ 500mL (from a primary or secondary thoracentesis, yielding in a high volume of tumor cells) for immunotherapy manufacture.
7. Tumor intended for immunotherapy manufacture is not embedded in bone and does not contain luminal tissue (e.g. bowel, ureter, bile duct).
8. Ability to understand and the willingness to sign a written protocol specific informed consent for tissue harvest or a parental/guardian informed consent and pediatric assent when appropriate.

Tissue Procurement Exclusion Criteria:

1. Medical condition requiring any form of chronic systemic immunosuppressive therapy (steroid or other) except physiologic replacement doses of hydrocortisone or equivalent (no more than 30 mg hydrocortisone or 10 mg prednisone equivalent daily) for < 30 days duration.
2. Known history of other malignancy unless having undergone curative intent therapy without evidence of that disease for ≥ 3 years except cutaneous squamous cell and basal cell skin cancer, superficial bladder cancer, in situ cervical cancer or other in situ cancers are allowed if definitively resected.
3. Brain metastases unless treated with curative intent (gamma knife or surgical resection) and without evidence of progression for ≥ 2 months.
4. Any documented history of autoimmune disease with exception of Type 1 diabetes on stable insulin regimen, hypothyroidism on stable dose of replacement thyroid medication, vitiligo, or asthma not requiring systemic steroids.
5. Known HIV or chronic Hepatitis B or C infection.
6. Known hypersensitivity to any temozolomide component or to dacarbazine (DTIC).
7. Known hypersensitivity to irinotecan or its excipients.
8. Known history of allergies or sensitivities to gentamicin.
9. History of or current evidence of any condition (including medical, psychiatric or substance abuse disorder), therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.

Study Enrollment Inclusion Criteria:

1. Completed manufacture of at least 4 vials of Vigil.
2. Karnofsky performance status (KPS) / Lansky performance status (LS) ≥80 percent.
3. Normal organ and marrow function as defined below:

   Absolute granulocyte count ≥1,000/mm3, Absolute lymphocyte count ≥400/mm3, Platelets ≥75,000/mm3, Hemoglobin ≥ 8.0 mg/dL, Total bilirubin ≤ institutional upper limit of normal*, AST(SGOT)/ALT(SGPT) ≤2x institutional upper limit of normal, Creatinine <1.5 mg/dL

   * documented Gilbert's syndrome may be considered after medical monitor review
4. Subject has recovered to CTCAE Grade 1 (except for parameters noted in Item 3, above) or better from all adverse events associated with prior therapy or surgery. Pre-existing motor or sensory neurologic pathology or symptoms, or dermatologic must be recovered to CTCAE Grade 2 or better.
5. If female of childbearing potential, has a negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a negative serum test will be required for study entry.
6. Ability to understand and the willingness to sign a written informed protocol specific consent or a parental/guardian informed consent and pediatric assent when appropriate.

Study Enrollment Exclusion Criteria:

In addition to the procurement exclusion criteria, subjects will NOT be eligible for study registration and randomization if meeting any of the following additional criteria:

1. Any anti-neoplastic therapy between tissue procurement for Vigil manufacture and start of study therapy.
2. Live vaccine used for the prevention of infectious disease administered < 30 days prior to the start of study therapy.
3. Post-surgery complication that in the opinion of the treating investigator would interfere with the patient's study participation or make it not in the best interest of the patient to participate.

Inclusion Criteria for Cross-Over:

Group B subjects will be eligible for cross-over, if they meet all of the following criteria:

1. Evidence of radiologic disease progression by RECIST 1.1 after enrollment into Group B.
2. Successful manufacturing of at least 4 vials of Vigil.
3. Karnofsky performance status (KPS) / Lansky performance status (LS) ≥70%.
4. Normal organ and marrow function as defined below:

   Absolute granulocyte count ≥1,000/mm3 Absolute lymphocyte count ≥400/mm3 Platelets ≥75,000/mm3 Total bilirubin ≤ institutional upper limit of normal AST(SGOT)/ALT(SGPT) ≤2x institutional upper limit of normal Creatinine <1.5 mg/dL

   *documented Gilbert's syndrome may be considered after medical monitor review.
5. Subject has recovered to CTCAE Grade 1 (except for parameters noted in Item 4, above) or better from all adverse events associated with prior therapy or surgery. Preexisting motor, sensory neurologic pathology or symptoms, or dermatologic toxicities must be recovered to CTCAE Grade 2 or better.
6. If female of childbearing potential, has a negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a negative serum test will be required for study entry.
7. Ability to understand and the willingness to sign a written informed protocol specific consent or a parental/guardian informed consent and pediatric assent when appropriate.

Exclusion Criteria for Cross-Over:

In addition to the Procurement and Study Enrollment exclusion criteria, Subjects will not be eligible for cross-over if meeting any of the following criteria:

1. With the exception of irinotecan and temozolomide while on study, any anti-neoplastic therapy between tissue procurement for Vigil manufacture and start of study therapy.
2. Live vaccine used for the prevention of infectious disease administered < 30 days prior to the start of study therapy.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Nemunaitis, MD, Study Director — Gradalis, Inc.
Locations (15):
- United States (15):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Los Angeles, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Dana-Farber/Boston Children's Cancer and Blood Disorders, Boston, Massachusetts
  - Washington University Siteman Cancer Center, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke Children's Hospital and Health Center; Duke Cancer Institute, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Texas Oncology - Pediatrics, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghisoli M, Rutledge M, Stephens PJ, Mennel R, Barve M, Manley M, Oliai BR, Murphy KM, Manning L, Gutierrez B, Rangadass P, Walker A, Wang Z, Rao D, Adams N, Wallraven G, Senzer N, Nemunaitis J. Case Report: Immune-mediated Complete Response in a Patient With Recurrent Advanced Ewing Sarcoma (EWS) After Vigil Immunotherapy. J Pediatr Hematol Oncol. 2017 May;39(4):e183-e186. doi: 10.1097/MPH.0000000000000822. PMID 28338569
- [Background] Ghisoli M, Barve M, Mennel R, Lenarsky C, Horvath S, Wallraven G, Pappen BO, Whiting S, Rao D, Senzer N, Nemunaitis J. Three-year Follow up of GMCSF/bi-shRNA(furin) DNA-transfected Autologous Tumor Immunotherapy (Vigil) in Metastatic Advanced Ewing's Sarcoma. Mol Ther. 2016 Aug;24(8):1478-83. doi: 10.1038/mt.2016.86. Epub 2016 Apr 25. PMID 27109631
- [Background] Ghisoli M, Barve M, Schneider R, Mennel R, Lenarsky C, Wallraven G, Pappen BO, LaNoue J, Kumar P, Nemunaitis D, Roth A, Nemunaitis J, Whiting S, Senzer N, Fletcher FA, Nemunaitis J. Pilot Trial of FANG Immunotherapy in Ewing's Sarcoma. Mol Ther. 2015 Jun;23(6):1103-1109. doi: 10.1038/mt.2015.43. Epub 2015 Mar 19. PMID 25917459
- [Background] Senzer N, Barve M, Kuhn J, Melnyk A, Beitsch P, Lazar M, Lifshitz S, Magee M, Oh J, Mill SW, Bedell C, Higgs C, Kumar P, Yu Y, Norvell F, Phalon C, Taquet N, Rao DD, Wang Z, Jay CM, Pappen BO, Wallraven G, Brunicardi FC, Shanahan DM, Maples PB, Nemunaitis J. Phase I trial of "bi-shRNAi(furin)/GMCSF DNA/autologous tumor cell" vaccine (FANG) in advanced cancer. Mol Ther. 2012 Mar;20(3):679-86. doi: 10.1038/mt.2011.269. Epub 2011 Dec 20. PMID 22186789

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirty-two (32) subjects signed consent for the tissue procurement portion of the study. Twenty-seven (27) subjects were not eligible to enroll into the main treatment portion of the study. Five (5) subjects were randomized into the main treatment portion of the study.
  Group B - crossover to receive 2nd Intervention with Vigil only:
  One (1) subject in Group B was not eligible to crossover to receive treatment with Vigil and 1 subject from Group B crossed over to receive Vigil.
Groups:
- Group A: Vigil in Combination With Irinotecan and Temozolomide: Participants randomized to Group A received oral temozolomide 100 mg/m2 daily (Days 1-5), total dose 500 mg/m2/cycle) and oral irinotecan 50 mg/m2 daily (Days 1-5, total dose 250 mg/m2/cycle). Vigil immunotherapy was administered at a concentration of 1 X 10e6 cells/dose given via intradermal injection on Day 15 of each cycle. 1 cycle = 21 days
  Participants continued treatment for a maximum of 12 cycles, or until disease progression, unacceptable toxicity, withdrawal of consent or other criterion is met for discontinuation from study.
Period: Main Study
Arm/Group | Group A: Vigil in Combination With Irinotecan and Temozolomide | Group B: Irinotecan and Temozolomide
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0
Period: Group B Crossover to Vigil Alone
Arm/Group | Group A: Vigil in Combination With Irinotecan and Temozolomide | Group B: Irinotecan and Temozolomide
Started | 0 (Crossover is not applicable to Group A.) | 1 (Only one subject from Group B was eligible to Crossover to receive treatment with Vigil.)
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only 1 subject randomized to Group B was eligible to Cross-over to receive Vigil.
Groups:
- Group A: Vigil in Combination With Irinotecan and Temozolomide: Participants randomized to Group A received oral temozolomide 100 mg/m^2 daily (Days 1-5), total dose 500 mg/m^2/cycle) and oral irinotecan 50 mg/m^2 daily (Days 1-5, total dose 250 mg/m^2/cycle). Vigil immunotherapy was administered at a concentration of 1 X 10e6 cells/dose given via intradermal injection on Day 15 of each cycle. 1 cycle = 21 days
  Participants continued treatment for a maximum of 12 cycles, or until disease progression, unacceptable toxicity, withdrawal of consent or other criterion is met for discontinuation from study.
- Group B: Irinotecan and Temozolomide: Participants randomized to Group B received oral temozolomide 100 mg/m^2 daily (Days 1-5), total dose 500 mg/m^2/cycle) and oral irinotecan 50 mg/m^2 daily (Days 1-5, total dose 250 mg/m^2/cycle).
  1 cycle = 21 days
  Participants continued treatment for a maximum of 12 cycles, or until disease progression, unacceptable toxicity, withdrawal of consent or other criterion is met for discontinuation from study.
- Total: Total of all reporting groups
Arm/Group | Group A: Vigil in Combination With Irinotecan and Temozolomide | Group B: Irinotecan and Temozolomide | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 2
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5
Baseline Performance Status [Count of Participants; unit: Participants] — An assessment of Performance Status (PS) on the Karnofsky or Lansky scale is standard way of measuring the ability of cancer patients to perform ordinary tasks. The PS scores range from 0 to 100. A higher score means the patient is better able to carry out daily activities. The assessment is made by an investigator during the physical exam of the subject.
  Participants
    80 | 0 | 2 | 2
    100 | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival (PFS) is defined as the time from randomization to the event of disease recurrence/progression according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria (version 1.1) for target lesions and assessed CT/MRI by local investigator.
Time Frame: From date of randomization until the date of first documented progression (assessed up to 3 years).
Population: PFS is not adequately assessable for difference between cohorts given only 5 participants were enrolled and received treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group A: Vigil in Combination With Irinotecan and Temozolomide | Group B: Irinotecan and Temozolomide
Number analyzed (Participants) | 3 | 2
Months | 2.8 [2.7 to NA] — N/A = Not Available. Upper confidence interval could not be calculated as there were insufficient number of participants with event. | 9.1 [2.8 to NA] — N/A = Not Available. Upper confidence interval could not be calculated as there were insufficient number of participants with event.

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as time from randomization to death or to the date of last follow-up. The date of last follow-up confirming survival will be used as the censoring date for subjects who are alive and/or do not have a known date of death.
Time Frame: From date of randomization until date of death from any cause, whichever came first (assessed up to 3 years).
Population: OS is not adequately assessable for difference between cohorts given only 5 participants were enrolled and received treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group A: Vigil in Combination With Irinotecan and Temozolomide | Group B: Irinotecan and Temozolomide
Number analyzed (Participants) | 3 | 2
Months | 16.1 [14.6 to NA] — N/A = Not Available. Upper confidence interval could not be calculated as there were insufficient number of participants with event. | 3.3 [3.3 to NA] — N/A = Not Available. Upper confidence interval could not be calculated as there were insufficient number of participants with event.

3. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the proportion of participants who have prolonged stable disease or a partial or complete response or complete response to therapy according to RECIST 1.1.
Time Frame: 6 months after treatment with Vigil.
Population: No subjects on trial achieved a partial or complete response, therefore the ORR was not determined.
Measure: Number; unit: Proportion of participants.
Arm/Group | Group A: Vigil in Combination With Irinotecan and Temozolomide | Group B: Irinotecan and Temozolomide
Number analyzed (Participants) | 3 | 2
Proportion of participants. | 0 | 0

4. Secondary Outcome: Vigil Manufacture Success Rate: Number of Participants Eligible for Treatment on the Main Study.
Description: Participants were considered eligible for treatment, if the tissue submitted to Gradalis met all criteria, including manufacturing product release criteria.
Time Frame: From manufacturing start date until 4 weeks post manufacturing for each tissue procurement (assessed up to 17 months).
Population: All enrolled subjects who completed tissue procurement and the tissue was received by Gradalis for Vigil Manufacture. Any subjects whose tissue was not submitted to Gradalis was excluded in the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Total Number of Tissue Procurements: Participants who underwent tissue procurement and the processed tissue samples were successfully shipped to Gradalis whereby Vigil production was attempted.
Arm/Group | Total Number of Tissue Procurements
Number analyzed (Participants) | 30
Participants | 4

ADVERSE EVENTS:
Time Frame: SAEs and Other Adverse Events: following procurement of the subject's tissue for tissue manufacture and for up to 30 days following the last study treatment, a duration of approximately 12 months. All-cause Mortality: from randomization date and until death or protocol termination, up to 3 years.
Description: All treated participants.
Groups:
- Group A: Vigil in Combination With Irinotecan and Temozolomide: Participants randomized to Group A received oral temozolomide 100 mg/m2 daily (Days 1-5), total dose 500 mg/m2/cycle) and oral irinotecan 50 mg/m2 daily (Days 1-5, total dose 250 mg/m2/cycle). Vigil immunotherapy was administered at a concentration of 1 X 10e6 cells/dose given via intradermal injection on Day 15 of each cycle. 1 cycle = 21 days
  Participants continued treatment for a maximum of 12 cycles, or until disease progression, unacceptable toxicity, withdrawal of consent or other criterion was met for discontinuation from study.
- Group B: Irinotecan and Temozolomide: Participants randomized to Group B received oral temozolomide 100 mg/m2 daily (Days 1-5), total dose 500 mg/m2/cycle) and oral irinotecan 50 mg/m2 daily (Days 1-5, total dose 250 mg/m2/cycle).
  1 cycle = 21 days
  Participants continued treatment for a maximum of 12 cycles, or until disease progression, unacceptable toxicity, withdrawal of consent or other criterion was met for discontinuation from study.
- Cross-over to Vigil Alone: Participants assigned to Group B crossed-over to received Vigil monotherapy at a concentration of 1 X 10e6 cells//dose via intradermal injection every 21 days following End of Treatment assessment.
  Participants received up to 12 doses of Vigil depending upon the quantity of Vigil manufactured.
Arm/Group | Group A: Vigil in Combination With Irinotecan and Temozolomide | Group B: Irinotecan and Temozolomide | Cross-over to Vigil Alone
All-Cause Mortality (participants affected / at risk) | 2/3 | 1/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/2 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Vigil in Combination With Irinotecan and Temozolomide (N=3) | Group B: Irinotecan and Temozolomide (N=2) | Cross-over to Vigil Alone (N=1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Vigil in Combination With Irinotecan and Temozolomide (N=3) | Group B: Irinotecan and Temozolomide (N=2) | Cross-over to Vigil Alone (N=1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (10) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (15) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Reflux esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 2 (7) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (8) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (2) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
ALT increased (Investigations) | 0 (0) | 1 (3) | 0 (0)
AST increased (Investigations) | 0 (0) | 1 (4) | 0 (0)
Bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Chloride increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hemoglobin increased (Investigations) | 0 (0) | 1 (5) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (5) | 0 (0)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (3) | 0 (0)
Platelets decreased (Investigations) | 0 (0) | 1 (4) | 0 (0)
WBC decreased (Investigations) | 0 (0) | 1 (8) | 1 (2)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (6) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ejaculation disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination of trial leading to small numbers of subjects analyzed. Technical problems with measurement leading to unreliable or uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT03495921/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/21/NCT03495921/SAP_001.pdf